CLINICAL TRIAL: NCT00559767
Title: Mapping of End Stage Renal Disease Genetic Susceptibility in African Americans by Admixture Linkage Disequilibrium
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906210; 06-C-N210
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Kidney Function; Genes; Association Analysis; Polymorphisms; Diabetes
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus

SUMMARY:
This study will identify which regions on the genes, and genes themselves, may account for an increased risk of end stage renal disease (ESRD), that is, near-total loss of kidney function, for people of African American descent. Researchers will use a technique called admixture linkage disequilibrium (MALD) to study genomes, genetic material, in about 2,500 participants from two existing studies and participants who will serve as controls. ESRD disproportionately affects African Americans, who constitute 29% of all ESRD patients in the Medicare ESRD program. The disease can result from a variety of diseases, with diabetes as the leading underlying cause (44% of cases) and hypertension as the second leading cause (26%). The proportion of ESRD cases caused by diabetes has increased dramatically.

Patients age 18 and older who are African American, who have ESRD, and who are participants of the FIND and CHOICE studies may be eligible for this study. FIND, or Family Investigation of Diabetes and Nephropathy, involves a multicenter study to identify susceptibility genes, that is, those with a risk, for diabetic and other forms of kidney disease. CHOICE, or Choices for Healthy Outcomes in Caring for ESRD patients is an ongoing study that identifies risk factors for cardiovascular outcomes in ESRD patients. The principle of mapping by MALD involves genetic variations that exist across populations. When mixing occurs between populations having different (heterogeneous) genes, the admixed offspring inherits chromosomes of distinct ancestry. However, over generations of mating, and recombination over several generations, originally large blocks of DNA from African ancestry have become part of smaller segments throughout the chromosome. The study will focus on risk alleles, that is, alternative forms of genes that carry a disease risk. Risk alleles are closely related to nearby ancestral gene markers found in a person.

Patients will undergo a collection of blood and urine for genetic testing. Researchers are conducting separate analyses in this study. Case-control analysis of ESRD will consist of 1,150 participants from FIND and 250 from CHOICE. There will also be 750 control participants from FIND. For the case-control analysis of diabetic ESRD, there will be about 750 participants from FIND, 125 from CHOICE, and 750 controls from FIND. Finally, there is the quantitative trait analysis, which looks at the phenotype-meaning visible characteristics produced by the interaction of a person's genetic makeup with the environment. That analysis will involve 350 patients with diabetic nephropathy but not ESRD and 750 controls from FIND.

DETAILED DESCRIPTION:
Background:

* End stage renal disease (ESRD) is the near-total loss of kidney function which can result from a variety of diseases. ESRD disproportionately affects African Americans; this group comprises 29% of all ESRD patients treated in the Medicare ESRD program, a proportion that markedly exceeds their representation in the general population.
* The Family Investigation of Diabetes and Nephropathy (FIND) study is an ongoing study to identify susceptibility genes for diabetic and other forms of nephropathy, and the Choices for Healthy Outcomes in Caring for ESRD patients (CHOICE) study is an ongoing prospective study to identify risk factors for cardiovascular outcomes in ESRD patients. Participants of these studies have already been recruited and characterized with respect to renal phenotypes; furthermore, DNAs from these individuals have already been collected and isolated. In this study, we intend to genotype markers suitable for MALD analysis in African Americans. The central hypothesis of the present study is that some renal disease susceptibility alleles are present at higher frequency in African Americans than in whites and that specific regions of the genome in African Americans contain marker alleles that are in admixture linkage disequilibrium with ESRD susceptibility alleles.

Objectives:

* The overall objective of this study is to identify novel loci, genes, and gene products, that may partially account for excess risk of end stage renal disease (ESRD) in African Americans compared to whites.
* To achieve this goal, we will employ Mapping by Admixture Linkage Disequilibrium (MALD) analysis, a specialized form of linkage disequilibrium mapping, to perform a genome-wide association study in approximately 2,500 African-American participants from the FIND and CHOICE studies.

Eligibility:

* Specific Inclusion/Exclusion criteria: African American
* Gender and minority inclusion. The FIND and CHOICE studies are open to both men and women of any ethnicity; however, due to the underlying principle of MALD analysis, this study will only include African-American participants of these cohorts.

Design:

* Genotype 1536 African-American MALD markers (2 cM average spacing) utilizing DNA from approximately 2,500 African-American participants in FIND and CHOICE.
* Perform a genome-wide association analysis utilizing a 2 cM dense genetic map and identify chromosomal loci that are in admixture linkage disequilibrium with:

  * ESRD in a case-control design
  * ESRD attributable to diabetes in a case-control design
  * Quantitative renal phenotypes
* Fine map putative chromosomal region in admixture linkage disequilibrium with ESRD with densely-spaced single nucleotide polymorphisms.
* A characterization of the MYH9 gene, its mRNA and the proteins encoded is planned for cases and controls. Gene sequencing of the region implicated will be undertaken. Characterization of mRNA products for quantities and alternative splicing will be evaluated. Experimental characterization of the MYH9 proteins for isoforms, post-translational modifications, interactions, and immunohistochemical staining will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA:

The cohorts utilized in this study, FIND and CHOICE, are open to adults of both genders and any ethnicity. However, we will select and utilize only those samples from African - American participants. We will also utilize African (Yorban) and European controls for genotyping from the NIGMS HGCR.

EXCLUSION CRITERIA:

Children and all ethnicities other than African - American, African, and European will be excluded from this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2860 (Estimated)
Dates: Start 2006-06-30; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Martha Linet, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Patterson N, Hattangadi N, Lane B, Lohmueller KE, Hafler DA, Oksenberg JR, Hauser SL, Smith MW, O'Brien SJ, Altshuler D, Daly MJ, Reich D. Methods for high-density admixture mapping of disease genes. Am J Hum Genet. 2004 May;74(5):979-1000. doi: 10.1086/420871. Epub 2004 Apr 14. PMID 15088269
- [Background] Smith MW, Patterson N, Lautenberger JA, Truelove AL, McDonald GJ, Waliszewska A, Kessing BD, Malasky MJ, Scafe C, Le E, De Jager PL, Mignault AA, Yi Z, De The G, Essex M, Sankale JL, Moore JH, Poku K, Phair JP, Goedert JJ, Vlahov D, Williams SM, Tishkoff SA, Winkler CA, De La Vega FM, Woodage T, Sninsky JJ, Hafler DA, Altshuler D, Gilbert DA, O'Brien SJ, Reich D. A high-density admixture map for disease gene discovery in african americans. Am J Hum Genet. 2004 May;74(5):1001-13. doi: 10.1086/420856. Epub 2004 Apr 14. PMID 15088270
- [Background] Smith MW, Lautenberger JA, Shin HD, Chretien JP, Shrestha S, Gilbert DA, O'Brien SJ. Markers for mapping by admixture linkage disequilibrium in African American and Hispanic populations. Am J Hum Genet. 2001 Nov;69(5):1080-94. doi: 10.1086/323922. PMID 11590548